CLINICAL TRIAL: NCT01407367
Title: Does Under-recognition of Kidney Disease Affect Patient Safety?
Brief Title: Safe Kidney Care Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey Fink, Associate Professor, Nephrology, University of Maryland, Baltimore
Other Study IDs: HP-00048532; R01DK084017 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-08-02 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Chronic Kidney Disease
Keywords: patient safety; chronic kidney disease; medical errors
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At each yearly research clinic visit (up to 4), 30 cc (6 teaspoons) of blood will be processed and stored for future assays related to kidney function.
  At first research clinic visit, 9 cc urine will be processed and stored for future assays related to kidney function.
  At each yearly research clinic visit, 1 swab of both nares, 1 pharyngeal swab and 1 skin swab will be obtained, processed and stored with future testing for multiple antibiotic resistant (MAR) organisms.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phase I and Phase II: Phase I (First 100 participants):
  Medical alert bracelet/necklace, Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
  Phase II (Next 250 participants):
  Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs

SUMMARY:
Chronic kidney disease (CKD) is common, but it is often over-looked in patients with this disease when they are getting medical treatment. Patients with CKD have special needs for their medical treatment. When these special needs are not considered their medical care may lead to unintended harm (called safety events) which can cause hospitalization, more kidney problems, and even death.

This research study has two purposes. The first purpose is to determine how participants feel about wearing a medical alert bracelet or necklace that alerts health care workers that the user of the bracelet or necklace has decreased kidney function. Medical alert bracelets are often recommended for people who have other medical problems, such as diabetes. This medical alert bracelet or necklace has an address to an informational website about the safe care of patients with kidney problems. The investigators think that alerting health care workers that a person has decreased kidney function may decrease their chances of having a medical injury and improve the safety of their care.

The second purpose of this research study is to track how often people with kidney problems may be exposed to medicines, tests, or procedures that might increase their chance of having an accidental medical injury or safety event. Though some medical injuries can not be prevented, the investigators want to find out what medical events in patients with kidney problems might be preventable. The investigators also want to find out if other things might increase a patient's chances of getting a medical injury, such as physical weakness or medical instructions that might be confusing.

DETAILED DESCRIPTION:
Chronic kidney disease not requiring dialysis (CKD) is common, but under-recognized, among patients who frequent the health care system, where improving patient safety is a high priority. Poor recognition of the disease and several other features unique to CKD make it a high-risk condition for adverse, patient-safety incidents (PSIs). In this context, PSIs refer to events of unintended harm or injury related to medications or medical care. These adverse safety events may include those usually cited for the general population (PSI), but also, CKD-specific unsafe practices (CKD-PSI) all of which, in turn, can lead to frequent hospitalization, accelerated loss of kidney function, increased risk of end-stage renal disease (ESRD), and death - all common outcomes in CKD. CKD-PSIs have been established in prior work by the investigators of this study with the help of an expert panel but it is not known how commonly PSIs or CKD-PSIs occur or how to measure these reliably in the CKD population. Furthermore, it is not known what role poor disease recognition plays in the occurrence of such safety events. Finally, it remains to be determined whether CKD-PSIs contribute to the high frequency of adverse outcomes so common in this disease. If CKD-PSIs are common and account for a significant portion of the adverse events so common in this population, then it is possible that by reducing the incidence of CKD-PSIs, through increased disease recognition, outcomes can be improved in this patient population.

In this study, the investigators will enroll volunteers from the population with pre-dialysis CKD for the purpose of observing the frequency of CKD-PSI in the target population detected over time. The participants will be assessed annually for events that relate to CKD-PSI. The first 100 participants (Phase I) will be provided with a standard medical alert accessory (bracelet or necklace) which is commonly used to alert doctors and other providers of a patient's disease state. In this case the medical alert accessory will state "Decreased Kidney Function. For My Care, Please Visit (website) www.safekidneycare.org" Participants are asked to log onto the website using unique 4-digit identifier (ID) assigned by the PI to track the participant's use of the website and to further improve the website. Since all information on the website is available to the public, participants are not required to use the ID to access the content of the website. The website does not collect or store patient health information, except for the Internet Protocol (IP) address which provides limited information on the location of the computer used to access the website (city, state, zip, and area code).

The volunteers in Phase I will be tracked over time as to whether they use and tolerate this medical alert bracelet/necklace and for their incidence of CKD-PSI. Enrollment will continue after Phase I in Phase II (n = 250) with participants tracked on an identical study schedule for detection of CKD-PSI. All study procedures are the same for Phase II except for the medical alert accessory. The overall goal of this study will be to determine: the frequency of CKD-PSI in the target population, the acceptability of an alert device (Phase I only) intended to increase the recognition of CKD, and the contribution of CKD-PSI to the high incidence of adverse outcomes in CKD

ELIGIBILITY:
Inclusion Criteria:

* estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2 (using Modified Diet in Renal Disease (MDRD) equation) based on the 2 out-patient serum creatinines obtained within the last 18 months and at least 90 days apart

Exclusion Criteria:

* <21 years of age,
* Expected to need dialysis within 12 months after time of enrollment,
* Expected to die within 12 months after time of enrollment,
* Unable to provide informed consent, or is a
* Prisoner
* Skin sensitivity or allergy to stainless steel and sterling silver (Phase 1 only)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a variety of chronic kidney disease (CKD) management and primary care setting. Some participants will be self-referrals.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Fink, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland Medical System, Baltimore, Maryland

REFERENCES:
- [Derived] Belkin MD, Doerfler RM, Wagner LA, Zhan M, Fink JC. Associations of Performance-Based Functional Assessments and Adverse Outcomes in CKD. Kidney360. 2021 Jan 19;2(4):629-638. doi: 10.34067/KID.0005802020. eCollection 2021 Apr 29. PMID 35373040
- [Derived] Diamantidis CJ, Fink W, Yang S, Zuckerman MR, Ginsberg J, Hu P, Xiao Y, Fink JC. Directed use of the internet for health information by patients with chronic kidney disease: prospective cohort study. J Med Internet Res. 2013 Nov 15;15(11):e251. doi: 10.2196/jmir.2848. PMID 24240617

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Phase I (first 108 participants enrolled) Medical alert bracelet/necklace, Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
- Phase II: Phase II (subsequent 242 participants enrolled) Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 108 | 242
Completed | 68 | 164
Not Completed | 40 | 78
Not completed — Death | 24 | 32
Not completed — Renal Replacement Therapy (RRT) | 12 | 29
Not completed — Withdrawal by Subject | 4 | 15
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Phase I (first 108 participants enrolled):
  Medical alert bracelet/necklace, Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
- Phase II: Phase II (subsequent 242 participants enrolled):
  Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 108 | 242 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 90 | 146
  >=65 years | 52 | 152 | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 61 | 99
  Male | 70 | 181 | 251
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 165 | 243
  White | 30 | 72 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 242 | 350
eGFR [Count of Participants; unit: Participants] — Estimated Glomerular Filtration Rate (eGFR) mL/min/1.73 m², baseline measure of kidney function, Stage 5 being the most severe stage of CKD (prior to ESRD) and Stage 2 being the most mild stage of CKD.
  Participants
    Stage 2 (60 ≤ eGFR ≤ 89 mL/min/1.73 m²) | 12 | 23 | 35
    Stage 3a (45 ≤ eGFR ≤ 59 mL/min/1.73 m²,) | 32 | 83 | 115
    Stage 3b (30 ≤ eGFR ≤ 44 mL/min/1.73 m²,) | 46 | 91 | 137
    Stage 4 (15 ≤ eGFR ≤ 29 mL/min/1.73 m²,) | 15 | 35 | 50
    Stage 5 (eGFR< 15 mL/min/1.73 m²,) | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Discrete Incidence of Any of the Chronic Kidney Disease Patient Safety Indicators (CKD-PSIs) Endorsed by the Consensus Expert Panel
Description: The discrete incidence of any of the following CKD-PSIs endorsed by the consensus expert panel:
  Class I events: Incidence of patient reported adverse events related to medical care or medicines incuding: Falling, Bleeding, Edema, Angioedema, Confusion or altered mental status, Rhabdomyolysis
  Class II events: Incidence of adverse events detected at annual study visits such as: Hyperkalemia, Hypokalemia, Hypoglycemia, Hyperglycemia, Orthostatic Hypotension, Hypotension, Hypertension, Bradycardia
  Class III events: Incidence of usage of medications or agents to be avoided in CKD and Incidence of improperly dosed medications in CKD
Time Frame: at the end of study (up to 4.25 years, depending on participant enrollment date)
Population: Safety events reported in this outcome measure are from 6 months prior to participant's annual in-center visits
Measure: Number; unit: events per 100 patient-visits
Groups:
- Phase I: Phase I Phase I (first 108 participants enrolled) Medical alert bracelet/necklace, Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
- Phase II: Phase II Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 108 | 242
events per 100 patient-visits
  Class I | 108.7 | 100.6
  Class II | 38.3 | 41.2

2. Secondary Outcome: Rate of All-cause Hospitalization
Description: Hospitalizations (following enrollment); including length of stay and safety events during hospitalization until time of end of study.
Time Frame: at the end of study (up to 4.25 years, depending on participant enrollment date)
Measure: Number; unit: events per patient-years
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 108 | 242
events per patient-years | 0.51 | 0.44

3. Secondary Outcome: Change in Renal Function From Baseline
Description: Renal function with estimated glomerular filtration rate (eGFR) based on serum creatinine measured annually until time of end of study.
Time Frame: at the end of study (up to 4.25 years, depending on participant enrollment date)
Measure: Median (Inter-Quartile Range); unit: ml/min per 1.73m^2 per month
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 108 | 242
ml/min per 1.73m^2 per month | -0.12 [-0.35 to 0.08] | -0.06 [-.38 to 0.16]

4. Secondary Outcome: Number of Participants With End-stage Renal Disease (ESRD) Defined as Need for Renal Replacement Therapy (Dialysis or Transplant)
Description: ESRD defined as the need for renal replacement therapy with either dialysis (hemodialysis or peritoneal) for 3 months or more; or renal transplantation up until the time of end of study.
Time Frame: at the end of study (up to 4.25 years, depending on participant enrollment date)
Measure: Number; unit: participants
Groups:
- Phase I: Phase I Medical alert bracelet/necklace, Medical event diary, Medical event ascertainment, Repeated measurement of renal function and other electrolytes, Review for CKD-PSIs
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 108 | 242
participants | 12 | 29
Statistical Analysis 1: Comparison: Phase I vs Phase II; Test type: Other; p = .04, Regression, Cox — calculated p-value. Results adjusted for gender, race, age, BMI, MAP, eGFR, smoking history, diabetes, hypertension, cardiovascular disease, cancer, education employment status, health literacy and RAAS use; Hazard Ratio (HR) = .38, 95% CI 2-sided [0.16 to 0.94]

5. Secondary Outcome: Number of Deaths Among Participants (All-cause)
Description: determined until end of study.
Time Frame: at the end of study (up to 4.25 years, depending on participant enrollment date)
Measure: Number; unit: participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 108 | 242
participants | 24 | 32
Statistical Analysis 1: Comparison: Phase I vs Phase II; Test type: Other; p = 0.86, Regression, Cox — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.53 to 1.99]

ADVERSE EVENTS:
Time Frame: up to 4.25 years, depending on participant enrollment date
Arm/Group | Phase I | Phase II
All-Cause Mortality (participants affected / at risk) | 24/108 | 32/242
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/242
Other Adverse Events (participants affected / at risk) | 0/108 | 0/242

LIMITATIONS AND CAVEATS:
Observational cohort with a sub-group to pilot a medical alert accessory; remainder of the cohort had no accessory. Bias cannot be excluded and direct group comparisons is not possible, nor can the accessory be formally evaluated as an intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT01407367/Prot_SAP_001.pdf